CLINICAL TRIAL: NCT01580488
Title: A Plaque Test Study With LEO 35299 in Psoriasis Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: PLQ-008; 2011-005349-11 (EudraCT Number)
Record Dates: First submitted 2012-04-16; First posted 2012-04-19 (Estimated); Results first posted 2013-12-30 (Estimated); Last update posted 2025-03-12 (Actual); Status verified 2013-11

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — Solutions

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: B LEO 35299 20 mg/g cream — once daily application, 3 weeks
Drug: C LEO 35299 20 mg/g cream — once daily application, 3 weeks
Drug: E LEO 35299 10 mg/g solution — once daily application, 3 weeks
Drug: F LEO 35299 10 mg/g solution — once daily application, 3 weeks
Drug: Daivonex® ointment — once daily application, 3 weeks
Drug: Daivonex® ointment vehicle — once daily application, 3 weeks

SUMMARY:
The purpose of the study is to evaluate the anti-psoriatic effect of LEO 35299 in different formulations, compared to Daivonex® ointment and Daivonex® ointment vehicle, using the psoriasis plaque test modified from the method developed by KJ Dumas and JR Scholtz.

ELIGIBILITY:
Inclusion Criteria:

1. Following verbal and written information about the trial, the subject must provide signed and dated informed consent before any study related activities are carried out.
2. Age 18 years or above.
3. Males, or females of non-child bearing potential.
4. Subjects with, in the opinion of the investigator, stable psoriasis based on Total Plaque Score evaluated at screening visit and at visit 2 (Baseline).

Exclusion Criteria:

1. Male subjects who are not willing to use a local contraception (such as condom) from the time of study entry and for three months following the last study drug application.
2. Female subjects who are pregnant, of child-bearing potential or who are breast feeding.
3. Systemic treatment with biological therapies (marketed or not marketed) with a possible effect on psoriasis vulgaris within 4 weeks (etanercept), 2 months(adalimumab, alefacept, infliximab), 4 months(ustekinumab) or 4 weeks/5 half-lives (which-ever islonger) for experimental biological products prior to randomisation and during the study.
4. Systemic treatments with all other therapies than biologicals, with a potential effect on psoriasis vulgaris (e.g., corticosteroids, retinoids, immune suppressants) within the 4-week period prior to randomisation and during the study.
5. Subjects using one of the following topical drugs for the treatment of psoriasis within the 4 week period prior to randomisation and during the study:

   - Potent or very potent (WHO group III-IV) corticosteroids.
6. Subjects using of phototherapy within the following time periods prior to randomisation and during the study:

   * PUVA (4 weeks)
   * UVB (2 weeks)
7. Subjects using one of the following topical drugs for the treatment of psoriasis within two weeks prior to randomisation and during the study:

   * WHO group I-II corticosteroids (except if used for treatment of scalp and/or facial psoriasis)
   * Topical retinoids
   * Vitamin D analogues
   * Topical immunomodulators (e.g. macrolides)
   * Anthracen derivatives
   * Tar,
   * Salicylic acid.
8. Subjects with current diagnosis of guttate, erythrodermic, exfoliative or pustular psoriasis
9. Subjects with known/suspected disorders of calcium metabolism associated with hypercalcemia within the last 10 years, based on medical history and/or subject interview
10. Subjects who have received treatment with any non-marketed drug substance (i.e., an agent which has not yet been made available for clinical use following registration) within the 4 week period prior to randomisation or longer, if the class of the substance requires a longer washout as defined above (e.g., biological treatments)
11. Subjects with current participation in any other interventional clinical, based on interview of the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Queille-Roussel, MD, Principal Investigator — Centre de Pharmacologie Clinique Appliquée à la Dermatologie (CPCAD), Hôpital l'Archet 2, 151 route Saint-Antoine de Ginestière 06202 Nice Cedex 3, France
Locations (1):
- Centre de Pharmacologie Clinique Appliquée à la Dermatologie (CPCAD) - Hôpital l'Archet 2, 151 route Saint-Antoine de Ginestière, Nice, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject first visit, start date: 24-Apr-2012 Last subject last visit, completion date: 05-Jun-2012
Pre-assignment Details: Prior to randomisation, the subjects entered a washout phase of up to 21 days (if required) where antipsoriatic treatment and other relevant medications or treatments had to be discontinued as defined by the exclusion criteria
Groups:
- All Study Participants: Each of the 24 subjects received all 6 investigational products on small dermal test sites: Topical cream formulation "B" containing 20 mg/g LEO 35299 Topical cream formulation "C" containing 20 mg/g LEO 35299 Topical solution formulation "E" containing 10 mg/g LEO 35299 Topical solution formulation "F" containing 10 mg/g LEO 35299 Topical ointment containing 50 mcg/g calcipotriol Topical ointment vehicle
Period: Overall Study
Arm/Group | All Study Participants
Started | 24
Completed | 23
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 19
Region of Enrollment [Number; unit: participants]
  France | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in the Total Clinical Score From Baseline to Day 22
Description: Investigator's rating of the clinical appearance of a psoriatic lesion. Maximum score is 9 (most severe); minimum score is 0 (least severe). The single items erythema, scaling, and infiltration (maximum score 3 each) are summed to obtain the Total Clinical Score. Total Clinical Score range from 0 (all symptoms absent) to 9 (all symptoms severe)
Time Frame: Baseline to Day 22
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- B LEO 35299 20 mg/g: Topical cream formulation "B" containing 20 mg/g LEO 35299
- C LEO 35299 20 mg/g: Topical cream formulation "C" containing 20 mg/g LEO 35299
- E LEO 35299 10 mg/g: Topical solution formulation "E" containing 10 mg/g LEO 35299
- F LEO 35299 10 mg/g: Topical solution formulation "F" containing 10 mg/g LEO 35299
- Daivonex® Ointment: Calcipotriol 50 mcg/g Ointment: Topical ointment containing 50 mcg/g calcipotriol
- Daivonex® Ointment: Topical ointment vehicle
Arm/Group | B LEO 35299 20 mg/g | C LEO 35299 20 mg/g | E LEO 35299 10 mg/g | F LEO 35299 10 mg/g | Daivonex® Ointment: Calcipotriol 50 mcg/g Ointment | Daivonex® Ointment
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
units on a scale | -2.8 (1.5) | -1.9 (1.5) | -1.5 (1.5) | -1.8 (1.7) | -4.0 (1.5) | -3.3 (1.5)

2. Secondary Outcome: Change in Erythema From Baseline to Day 22
Description: Investigator's rating of the clinical appearance of erythema. Maximum score is 3 (most severe); minimum score is 0 (absent).
Time Frame: Baseline to Day 22
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | B LEO 35299 20 mg/g | C LEO 35299 20 mg/g | E LEO 35299 10 mg/g | F LEO 35299 10 mg/g | Daivonex® Ointment: Calcipotriol 50 mcg/g Ointment | Daivonex® Ointment
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
units on a scale | -0.91 (0.56) | -0.67 (0.60) | -0.54 (0.47) | -0.70 (0.60) | -1.09 (0.56) | -1.07 (0.53)

3. Secondary Outcome: Change in Infiltration From Baseline to Day 22
Description: Investigator's rating of the clinical appearance of infiltration. Maximum score is 3 (most severe); minimum score is 0 (absent).
Time Frame: Baseline to Day 22
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | B LEO 35299 20 mg/g | C LEO 35299 20 mg/g | E LEO 35299 10 mg/g | F LEO 35299 10 mg/g | Daivonex® Ointment: Calcipotriol 50 mcg/g Ointment | Daivonex® Ointment
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
units on a scale | -0.87 (0.59) | -0.59 (0.54) | -0.46 (0.58) | -0.46 (0.66) | -1.48 (0.55) | -1.11 (0.54)

4. Secondary Outcome: Change in Scaling From Baseline to Day 22
Description: Investigator's rating of the clinical appearance of scaling . Maximum score is 3 (most severe); minimum score is 0 (absent).
Time Frame: Baseline to Day 22
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | B LEO 35299 20 mg/g | C LEO 35299 20 mg/g | E LEO 35299 10 mg/g | F LEO 35299 10 mg/g | Daivonex® Ointment: Calcipotriol 50 mcg/g Ointment | Daivonex® Ointment
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
units on a scale | -1.09 (0.49) | -0.74 (0.60) | -0.61 (0.64) | -0.67 (0.60) | -1.52 (0.59) | -1.30 (0.49)

5. Secondary Outcome: Change in Lesion Thickness From Baseline to Day 22
Description: Change in total skin thickness measured by ultrasound from baseline to end of treatment
Time Frame: Baseline to Day 22
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | B LEO 35299 20 mg/g | C LEO 35299 20 mg/g | E LEO 35299 10 mg/g | F LEO 35299 10 mg/g | Daivonex® Ointment: Calcipotriol 50 mcg/g Ointment | Daivonex® Ointment
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
millimeters | -0.31 (0.37) | -0.18 (0.31) | -0.22 (0.45) | -0.24 (0.33) | -0.36 (0.37) | -0.38 (0.36)

6. Secondary Outcome: Change in Skin Thickness From Baseline to Day 22
Description: Change in skin thickness - echo-poor band measured by ultrasound from baseline to end of treatment
Time Frame: Baseline to Day 22
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | B LEO 35299 20 mg/g | C LEO 35299 20 mg/g | E LEO 35299 10 mg/g | F LEO 35299 10 mg/g | Daivonex® Ointment: Calcipotriol 50 mcg/g Ointment | Daivonex® Ointment
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
millimeters | -0.40 (0.56) | -0.29 (0.47) | -0.24 (0.71) | -0.40 (0.51) | -0.57 (0.57) | -0.49 (0.35)

ADVERSE EVENTS:
Arm/Group | B LEO 35299 20 mg/g | C LEO 35299 20 mg/g | E LEO 35299 10 mg/g | F LEO 35299 10 mg/g | Daivonex® Ointment: Calcipotriol 50 mcg/g Ointment | Daivonex® Ointment
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24 | 2/24 | 1/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | B LEO 35299 20 mg/g (N=24) | C LEO 35299 20 mg/g (N=24) | E LEO 35299 10 mg/g (N=24) | F LEO 35299 10 mg/g (N=24) | Daivonex® Ointment: Calcipotriol 50 mcg/g Ointment (N=24) | Daivonex® Ointment (N=24)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1

LIMITATIONS AND CAVEATS:
This was an exploratory study in which each of the 24 subjects received all 6 treatments on 2 cm diameter dermal test sites. Regarding Adverse Events, only local dermal reactions could be potentially attributed to a specific treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor is entitled to review and comment on publications prior to submission or presentation. Upon request of the sponsor, the investigator shall delay publication or presentation to allow for protection of the sponsors inventions and other intellectual property.